CLINICAL TRIAL: NCT03407391
Title: Antecedents of Picky Eating Behaviour in Young Children
Brief Title: Antecedent Picky Eating Behaviour in Young Children
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry); Wellcome Trust (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: ALSPAC
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Child Behavior; Child Rearing; Eating Behavior; Parent-Child Relations; Parenting; Feeding and Eating Disorders of Childhood
Keywords: Picky eater; Fussy eater; Faddy eater; Nutrition
MeSH Terms: conditions — Child Behavior; Feeding Behavior; Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Picky eater: Identified as a very picky eater from parental questionnaire
  Interventions: Other: None - observational
- Not a picky eater: Identified as not a picky eater from parental questionnaire
  Interventions: Other: None - observational
- Somewhat picky eater: Identified as a somewhat picky eater from parental questionnaire
  Interventions: Other: None - observational

INTERVENTIONS:
Other: None - observational — No intervention - observational only

SUMMARY:
Picky eating behaviour in young children is a very common concern for parents. The aim of the study is to investigate factors during early life which are associated with a child becoming a picky eater.

DETAILED DESCRIPTION:
Singleton children from the Avon Longitudinal Study of Parents and Children will be studied prospectively (n=5758-6608). Parental-completion questionnaires will be used to define 'picky eating' status at age 3 years, and child and parental feeding behaviours and practices throughout the first 2 years of the child's life. Multinomial logistic regression models with 3 levels of picky eating status (not, somewhat and very picky) as the dependant variables will be used to test associations with antecedent variables, first assessing variables from pregnancy, and the first and second year of life, separately, then combining all significant variables in a final model.

ELIGIBILITY:
Inclusion Criteria:

* Child enrolled in ALSPAC, singleton, parent answered question on picky eating behaviour in questionnaire

Exclusion Criteria:

* Child not enrolled in ALSPAC, multiple, parent did not answer question on picky eating behaviour in questionnaire

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All pregnant women in the former Avon Health Authority with an expected delivery date between April 1991 and December 1992 were eligible for the study; 14,541 pregnant women were initially enrolled, resulting in a cohort of 14,062 live births with 13,988 alive at 1 year of age. Parents/caregivers were sent a questionnaire when the child was 3 years old that included a question on picky eating behaviour. Singleton children whose parents/caregivers answered this question were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 6608 (Actual)
Dates: Start 1991-04-01 (Actual); Primary Completion 1995-12-01 (Actual); Study Completion 1995-12-01 (Actual)

PRIMARY OUTCOMES:
Being a very picky eater or not at age 3 years | Age 3 years
  Parent/caregiver answers 'yes, very' or 'no' to question on picky eating in questionnaire

SECONDARY OUTCOMES:
Being a somewhat picky eater at age 3 years | Age 3 years
  Parent/caregiver answers 'somewhat' to question on picky eating in questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nic Timpson, PhD, Study Director — University of Bristol

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set — http://www.bristol.ac.uk/alspac/ — ALSPAC data is available for use by researchers on application through the website